CLINICAL TRIAL: NCT03250949
Title: Clinical Evaluation Of Dental Implants Stability Placed In Healed Bony Sites Following Over-drilling Compared To Conventional-Drilling Protocol: A Randomized Controlled Trial.
Brief Title: Clinical Evaluation Of Dental Implants Stability Placed In Healed Bony Sites Following Over-drilling Compared To Conventional-Drilling Protocol
Acronym: RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azhar ALI ELSAYED SELEEM (Other)
Responsible Party: Sponsor-Investigator, Azhar ALI ELSAYED SELEEM, doctor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Randomized Controlled Trial
Record Dates: First submitted 2017-08-10; First posted 2017-08-16 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Crestal Bone Resorption; Implant Primary Stability; Implant Osseointegration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional-Drilling Tight Fit (Control) group (No Intervention): osteotomy will be achieved with no. 6 round , then widened , using a drill 1 mm larger than the final drill provided by the manufacturer. the final size of the control osteotomies were same diameter of the implant.
- Over-drilling Loose Fit (Test) group (Experimental): Osteotomy preparations for the loose fit group will be identical to those of the tight fit group until final drill, which will be 0.2mm wider than the diameter of the implant.
  Interventions: Procedure: implant site over drilling protocol

INTERVENTIONS:
Procedure: implant site over drilling protocol — Osteotomy preparations for the loose fit group will be identical to those of the tight fit group until final drill, which will be 0.2mm wider than the diameter of the implant.
  osteotomy site of the implant is wider by 0.2mm than the implant diameter
  Other Names: NEO biotech implant system
  Arms: Over-drilling Loose Fit (Test) group

SUMMARY:
Clinical Evaluation Of Dental Implants Stability Placed In Healed Bony Sites Following Over-drilling Compared To Conventional-Drilling Protocol

DETAILED DESCRIPTION:
- Statement of the problem:

peri-implant bone is affected by excessive mechanical stress, the mechanism of bone formation is reduced and the bone resorption is increased, leading to MBL. Isidor F. 2006, Warreth A, 009 A drilling sequence using a drill that is smaller than the implant diameter has been applied as a way to obtain enough initial stability.Bilhan H,2010 However, the implant can be extremely compressed or exceed the torque, which can be higher than the elastic limit of bone when a drill that is smaller than the implant diameter is used. This may affect the bone surrounding the implant and may also lead to a micro fracture.

Frost mentioned that alveolar bone density is changed by micro deformation due to modification of the physical condition. Bone resorption and fibrous tissue production progress if the micro deformation rate is higher than 3,000 micro strain (με). Also, continuous bone replacement occurs while woven bone appears. Wolff J.1986 Bone tissue adapts to the change of stress while minimizing its weight and transforming its structure. Frost HM,1989 The bone formation mechanism is inhibited and the bone resorption mechanism is enhanced if excessive mechanical stress is applied to alveolar bone during implantation, resulting in the progression of marginal bone loss (MBL). Isidor F.2006 , Warreth A,2009-

Rationale for carrying out the trial:

Success and survival rate of an implant are directly associated with primary stability. Friberg B,et al 1991 Primary stability is achieved with initial rigid fixation of implants during the surgery and considered necessary for a successful osseointegration. Sennerby L,et al 1992, Rodrigo D,et al 2010 There are two different processes of bone formation at implant sites; contact and distance osteogenesis. Contact osteogenesis infers new bone formation in direct contact with the implant surface. Distance osteogenesis is the new bone formation on the surfaces of the parent bone and occurs when primary stability is absent at implant site. Davies JE.et al 2003, Sivolella S,et al2012

When there is a gap between the implant surface and bone, a clot will fill the space and will be replaced by a provisional connective matrix that will act as scaffold for formation of woven bone. Berglundh T,et al,2003 , Rossi F,2012 Our study will evaluate the effect of oversized drilling on implant success and secondary stability

ELIGIBILITY:
Inclusion Criteria:

* Patients who have at least one missing tooth in the upper maxillary arch.
* Patients with healthy systemic condition.(Brightman. 1994)
* Patients aged from 20 to 60 years old.
* Good oral hygiene.(Wiesner et al. 2010)
* Accepts 9 months follow-up period (cooperative patients)
* Patient provides an informed consent.

Exclusion Criteria:

* Patients with signs of acute infection related to the area of interest.
* Patients with habits that may jeopardize the implant longevity and affect the results of the study such as parafunctional habits (Lobbezoo et al. 2006).
* Current and former smokers (Lambert, Morris, and Ochi 2000)
* Pregnant women

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
implant stability | first 3 months
  Resonance frequency analysis (RFA) OSSTELL (Osstell Resonance frequency analysis (RFA) (Osstell

SECONDARY OUTCOMES:
Crestal bone level | from 3 to 6 month
  by Digital radiography